CLINICAL TRIAL: NCT07012265
Title: An Investigation of the Factors Related to Attitudes Towards Hospice and Palliative Care Among the Bunun Tribe in Taiwan: A Case Study of the Lona Village in Nantou
Brief Title: An Investigation of the Factors Related to Attitudes Towards Hospice and Palliative Care Among the Bunun Tribe in Taiwan
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Kwo-Chen Lee, Professor, China Medical University Hospital
Other Study IDs: CMUH113-REC3-127
Record Dates: First submitted 2025-04-28; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Resilience; Hospice Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The study plans to enroll 82 participants. Inclusion criteria include: 1) being twenty years of age or older; 2) residing in Lona Village, Xinyi Township, Nantou County for at least twenty years; 3) being literate with at least an elementary level of reading ability to complete structured questionnaires. Research instruments include the Faith Maturity Scale, Resilience Scale, and Attitudes Toward Hospice and Palliative Care Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to investigate the factors related to attitudes towards hospice and palliative care among the Bunun tribe in Taiwan, with a specific focus on the influence of faith maturity and resilience. A cross-sectional study will be conducted in Lona Village, Nantou County, enrolling 82 Bunun participants aged 20 and above, who have resided in the village for at least 20 years. Participants must possess basic literacy skills and will complete structured questionnaires assessing faith maturity, resilience, and attitudes towards hospice and palliative care. Pearson correlation tests will be used for data analysis, with significance set at p &lt; 0.05. The expected outcome is to provide empirical data on the relationship between faith maturity, resilience, and attitudes towards hospice care among the Bunun, contributing to healthcare policy tailored to Indigenous communities.

DETAILED DESCRIPTION:
The detailed design of this study emphasizes the cultural and spiritual dimensions that influence the Bunun tribe is attitudes toward hospice and palliative care. The Bunun tribe's cultural perspectives on death, illness, and caregiving differ from other ethnic groups in Taiwan. Faith plays a crucial role in the daily lives of the Bunun, while resilience reflects their capacity to cope with adversity, both of which may be key determinants of their attitudes toward hospice care.

Validated research instruments, such as the Faith Maturity Scale and Resilience Scale, are used to assess the participant is faith and psychological conditions. Additionally, the Attitudes Toward Hospice and Palliative Care Scale will help researchers gauge the level of acceptance and potential concerns regarding hospice care.

The cross-sectional design allows for the collection of sufficient data for an initial analysis to identify the relationship between faith maturity, resilience, and attitudes toward hospice care. Based on these findings, the research team will be able to provide specific recommendations to improve awareness and acceptance of hospice care among the Bunun and other Indigenous communities in Taiwan, thus contributing to more culturally appropriate healthcare service designs and policies.

ELIGIBILITY:
Inclusion Criteria:

Aged 20 years or older Resided in Lona Village, Xinyi Township, Nantou County for at least 20 years Literate with at least an elementary level of reading ability to complete structured questionnaires

Exclusion Criteria:

Individuals with hearing impairments or speech disorders Individuals diagnosed with emotional disorders by a physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) being twenty years of age or older; (2) residing in Lona Village, Xinyi Township, Nantou County for at least twenty years; (3) being literate with at least an elementary level of reading ability to complete structured questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Explore the current status and related factors of faith maturity, resilience, and attitudes towards hospice and palliative care among the Bunun tribe in Taiwan. | The plan is to collect structured questionnaire responses from 82 Bunun Indigenous people within three months.
  Structured questionnaires will be administered to 82 Bunun Indigenous adults to assess:
  1. Faith Maturity (FMS, score range: 12-84; higher = greater faith maturity)
  2. Resilience (RS-14, score range: 14-98; higher = greater resilience)
  3. Palliative Care Attitudes (score range: 20-100; higher = more favorable attitudes)

CONTACTS AND LOCATIONS:
Overall Officials: KwoChen Lee, ph.D, Study Director — 011+886+4+22053366#7102
Locations (1):
- Luona Village, Xinyi Township, Nantou City, Taiwan 556, Nantou City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoo SH, Kim M, Yun YH, Keam B, Kim YA, Kim YJ, Shim HJ, Song EK, Kang JH, Kwon JH, Lee JL, Lee SN, Kim SY, Kang EJ, Do YR, Choi YS, Jung KH. Attitudes toward early palliative care in cancer patients and caregivers: a Korean nationwide survey. Cancer Med. 2018 May;7(5):1784-1793. doi: 10.1002/cam4.1441. Epub 2018 Mar 25. PMID 29577624
- [Background] Tang ST, Huang EW, Liu TW, Wang HM, Chen JS. A population-based study on the determinants of hospice utilization in the last year of life for Taiwanese cancer decedents, 2001-2006. Psychooncology. 2010 Nov;19(11):1213-20. doi: 10.1002/pon.1690. PMID 20119936
- [Background] Tan WS, Beatty L, Koczwara B. Do cancer patients use the term resilience? A systematic review of qualitative studies. Support Care Cancer. 2019 Jan;27(1):43-56. doi: 10.1007/s00520-018-4456-y. Epub 2018 Sep 12. PMID 30209600
- [Background] Stewart DE, Yuen T. A systematic review of resilience in the physically ill. Psychosomatics. 2011 May-Jun;52(3):199-209. doi: 10.1016/j.psym.2011.01.036. PMID 21565591
- [Background] Spence ND, Wells S, Graham K, George J. Racial Discrimination, Cultural Resilience, and Stress. Can J Psychiatry. 2016 May;61(5):298-307. doi: 10.1177/0706743716638653. Epub 2016 Mar 28. PMID 27254805
- [Background] Polit DF, Beck CT, Owen SV. Is the CVI an acceptable indicator of content validity? Appraisal and recommendations. Res Nurs Health. 2007 Aug;30(4):459-67. doi: 10.1002/nur.20199. PMID 17654487
- [Background] Pandya SP. Faith Maturity and Mental Well-Being: A Longitudinal Study of Indian American Followers of a Guru Tradition. J Relig Health. 2020 Apr;59(2):743-757. doi: 10.1007/s10943-018-0632-0. PMID 29730808
- [Background] Ni K, Gong Y, Li F, Cao X, Zhang H, Chu H, Li T, Mairipaiti A, Zhao Y, Li N. Knowledge and attitudes regarding hospice care among outpatients and family members in two hospitals in China. Medicine (Baltimore). 2019 Apr;98(16):e15230. doi: 10.1097/MD.0000000000015230. PMID 31008953
- [Background] Narayan MC. Culture's effects on pain assessment and management. Am J Nurs. 2010 Apr;110(4):38-47; quiz 48-9. doi: 10.1097/01.NAJ.0000370157.33223.6d. PMID 20335689
- [Background] Min S. [The relationship between maturity of Christian faith and anxiety of patients with cancer]. Kanho Hakhoe Chi. 1989 Apr;19(1):118-26. doi: 10.4040/jnas.1989.19.1.118. Korean. PMID 2739232
- [Background] Maggi S, Roberts W, MacLennan D, D'Angiulli A. Community resilience, quality childcare, and preschoolers' mental health: a three-city comparison. Soc Sci Med. 2011 Oct;73(7):1080-7. doi: 10.1016/j.socscimed.2011.06.052. Epub 2011 Jul 22. PMID 21835523
- [Background] Lau J, Khoo AM, Ho AH, Tan KK. Psychological resilience among palliative patients with advanced cancer: A systematic review of definitions and associated factors. Psychooncology. 2021 Jul;30(7):1029-1040. doi: 10.1002/pon.5666. Epub 2021 Mar 16. PMID 33728728
- [Background] Jordan RI, Allsop MJ, ElMokhallalati Y, Jackson CE, Edwards HL, Chapman EJ, Deliens L, Bennett MI. Duration of palliative care before death in international routine practice: a systematic review and meta-analysis. BMC Med. 2020 Nov 26;18(1):368. doi: 10.1186/s12916-020-01829-x. PMID 33239021
- [Background] Hou CC, Kuo T. Home Care Services for Indigenous Population in Taiwan: Cultural and Socio-Structural Implications for Long-Term Care Policy. J Gerontol Soc Work. 2019 Apr;62(3):306-323. doi: 10.1080/01634372.2019.1575307. Epub 2019 Feb 11. PMID 30739607
- [Background] Hasson F, Nicholson E, Muldrew D, Bamidele O, Payne S, McIlfatrick S. International palliative care research priorities: A systematic review. BMC Palliat Care. 2020 Feb 3;19(1):16. doi: 10.1186/s12904-020-0520-8. PMID 32013949
- [Background] Gomez-Virseda C, de Maeseneer Y, Gastmans C. Relational autonomy in end-of-life care ethics: a contextualized approach to real-life complexities. BMC Med Ethics. 2020 Jun 30;21(1):50. doi: 10.1186/s12910-020-00495-1. PMID 32605569
- [Background] Fleming J, Ledogar RJ. Resilience and Indigenous Spirituality: A Literature Review. Pimatisiwin. 2008 Summer;6(2):47-64. PMID 20963185
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Choi JY, Chang YJ, Song HY, Jho HJ, Lee MK. Factors that affect quality of dying and death in terminal cancer patients on inpatient palliative care units: perspectives of bereaved family caregivers. J Pain Symptom Manage. 2013 Apr;45(4):735-45. doi: 10.1016/j.jpainsymman.2012.04.010. Epub 2012 Oct 25. PMID 23102560
- [Background] Chen C, Sun X, Liu Z, Jiao M, Wei W, Hu Y. The relationship between resilience and quality of life in advanced cancer survivors: multiple mediating effects of social support and spirituality. Front Public Health. 2023 Aug 28;11:1207097. doi: 10.3389/fpubh.2023.1207097. eCollection 2023. PMID 37701908
- [Background] An AR, Lee JK, Yun YH, Heo DS. Terminal cancer patients' and their primary caregivers' attitudes toward hospice/palliative care and their effects on actual utilization: A prospective cohort study. Palliat Med. 2014 Jul;28(7):976-985. doi: 10.1177/0269216314531312. Epub 2014 Apr 29. PMID 24781817
- [Background] Allen J, Hopper K, Wexler L, Kral M, Rasmus S, Nystad K. Mapping resilience pathways of Indigenous youth in five circumpolar communities. Transcult Psychiatry. 2014 Oct;51(5):601-31. doi: 10.1177/1363461513497232. Epub 2013 Aug 21. PMID 23965730
- See also: Religion and Health: Public Health Research and Practice — https://www.annualreviews.org/content/journals/10.1146/annurev.publhealth.21.1.335
- See also: Palliative care: patient's autonomy in the end-of-life situation — https://link.springer.com/article/10.1007/s12254-021-00783-5
- See also: The Pursuit of Resilience: A Meta-Analysis and Systematic Review of Resilience-Promoting Interventions — https://ideas.repec.org/a/spr/jhappi/v23y2022i4d10.1007_s10902-021-00452-8.html
- See also: Resilience Processes in Development: Fostering Positive Adaptation in the Context of Adversity. — https://awspntest.apa.org/record/2005-04216-002
- See also: Death, Emotions, and Social Change among the Austronesian-Speaking Bunun of Taiwan — https://repository.kulib.kyoto-u.ac.jp/dspace/bitstream/2433/152154/1/490203.pdf